CLINICAL TRIAL: NCT03239145
Title: Phase Ib Study to Test the Safety and Potential Synergy of Pembrolizumab (Anti-PD-1) and AMG386 (Angiopoietin-2 (Ang-2) in Patients With Advanced Solid Tumor
Brief Title: Pembrolizumab (Anti-PD-1) and AMG386 (Angiopoietin-2 (Ang-2) in Patients With Advanced Solid Tumor
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Amgen (Industry)
Responsible Party: Principal Investigator, F. Stephen Hodi, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-217
Record Dates: First submitted 2017-08-01; First posted 2017-08-03 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Advanced Solid Tumor
Keywords: Advanced Solid Tumor; Melanoma; Ovarian Cancer; Renal Cancer; Colorectal Cancer
MeSH Terms: conditions — Melanoma; Ovarian Neoplasms; Kidney Neoplasms; Colorectal Neoplasms | interventions — pembrolizumab; trebananib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Pembrolizumab + Trebananib (Experimental): Part 1 Standard 3+3 Dose Escalation
  Interventions: Drug: Pembrolizumab; Drug: Trebananib
- Pembrolizumab + Trebananib (Melanoma) (Experimental): Part 2 Dose Expansion
  Interventions: Drug: Pembrolizumab; Drug: Trebananib
- Pembrolizumab + Trebananib (Ovarian) (Experimental): Part 2 Dose Expansion
  Interventions: Drug: Pembrolizumab; Drug: Trebananib
- Pembrolizumab + Trebananib (Colorectal) (Experimental): Part 2 Dose Expansion
  Interventions: Drug: Pembrolizumab; Drug: Trebananib
- Pembrolizumab + Trebananib (Renal Cell Carcinoma) (Experimental): Part 2 Dose Expansion
  Interventions: Drug: Pembrolizumab; Drug: Trebananib

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab is designed to augment the natural ability of the immune system to recognize and target cancer cells
  Other Names: Keytruda
Drug: Trebananib — AMG386 is a drug that may kill tumor cells and blocks blood vessels that supply the tumor with nutrients and oxygen
  Other Names: AMG 386

SUMMARY:
This research study is studying an investigational combination of drugs as a possible treatment for advanced solid tumors: melanoma, ovarian, renal, or colorectal cancer.

The drugs involved in this study are:

* Pembrolizumab
* AMG386

DETAILED DESCRIPTION:
This research study is a Phase Ib clinical trial, which tests the safety of an investigational combination of drugs and also tries to define the appropriate dose of the investigational drugs to use for further studies. "Investigational" means that the drug is being studied.

FDA (the U.S. Food and Drug Administration) has not approved of the combination of the study drugs pembrolizumab and AMG386 as a treatment for any disease. However, the FDA has approved pembrolizumab by itself for melanoma and non-small cell lung cancer.

Pembrolizumab is a humanized monoclonal antibody, or specialized type of protein, produced in the laboratory for use in treating patients with the participant disease. Pembrolizumab is designed to augment the natural ability of the immune system to recognize and target cancer cells.

AMG386 is a drug that may kill tumor cells and blocks blood vessels that supply the tumor with nutrients and oxygen. Drugs that block blood vessel formation are called "anti-angiogenic" therapies. AMG386 has been used and is currently being used in other clinical trials treating different types of cancer. Information from these other clinical trials suggests that this drug may help stop tumor growth.

In this research study, the investigators are interested in looking at the combination of AMG386 with pembrolizumab because research done in the laboratory has suggested that the immunotherapy effect could be limited by the presence of tumor vessels in a process called angiogenesis. Adding AMG386 to pembrolizumab may help overcome this limitation and augment the effect of pembrolizumab.

This combination of study drugs is being researched to:

* Determine the safety and tolerability of pembrolizumab and AMG386 at different dose levels.
* Determine the side effects of pembrolizumab and AMG386 when they are given in combination
* Determine if pembrolizumab in combination with AMG386 is a possible treatment for cancer
* Determine if pembrolizumab in combination with AMG386 changes immune cells in the blood or tumor

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to provide written informed consent for the trial.
* Be ≥ 18 years of age on day of signing informed consent.
* Have measurable disease based on RECIST 1.1.
* In dose escalation (Phase I), patients must have histologically or cytologically confirmed metastatic disease from any solid tumor that is incurable and fulfills one of the following criteria:

  * Has demonstrated progression of disease following at least one line of effective systemic therapy. Prior treatment with anti-CTLA-4 antibody (including ipilimumab) is allowable OR
  * For which effective therapy does not exist
* In dose expansion (part 2), patients must have histologically or cytologically confirmed unresectable or metastatic melanoma, renal cell carcinoma, ovarian cancer, or colorectal cancer.
* Renal cell patients must have had at least one prior VEGF TKI.
* Ovarian cancer patients must be resistant to platinum therapy (i.e. within 6 months of last platinum therapy).
* Patients with colorectal cancer should have progressed on at least one fluorouracil plus irinotecan or oxaliplatin containing regimen.
* Patients with melanoma should have unresectable or metastatic disease. Melanoma patients with BRAF V600E or V600K mutation-positive melanoma who have previously received a BRAF inhibitor with or without a MEK inhibitor) are eligible.
* In the dose expansion cohort patients should be willing to provide tissue from a newly obtained core or excisional biopsy of a tumor lesion (pre-treatment) and post-treatment biopsy. Newly-obtained is defined as a specimen obtained up to 6 weeks (42 days) prior to initiation of treatment on Day 1. Patients for whom newly-obtained samples cannot be provided (e.g., inaccessible, subject safety concern, or unwilling to undergo biopsy) may submit an archived specimen only upon agreement from the Sponsor. An on-treatment biopsy will be collected approximately halfway through the induction period, about 6 weeks from the start of study treatment (sometime between Cycle 2 Day 8 - Cycle 3 Day 1).
* Have a performance status of 0 or 1 on the ECOG Performance Scale (see Appendix A) up to 28 days before treatment initiation
* Demonstrate adequate organ function as defined in Table 1, all screening labs should be performed up to 28 days before treatment initiation.
* System Laboratory Value
* Hematological

  * Absolute neutrophil count (ANC) ≥1,500 /mcL
  * Platelets ≥100,000 / mcL
  * Hemoglobin ≥9 g/dL or ≥5.6 mmol/L without transfusion or EPO dependency (within 7 days of assessment)
* Renal

  --Serum creatinine OR Measured or ≤1.5 X upper limit of normal (ULN) OR calculateda creatinine clearance ≥60 mL/min for subject with creatinine levels (GFR can also be used in place of > 1.5 X institutional ULN creatinine or CrCl)
* Hepatic

  * Serum total bilirubin ≤ 1.5 X ULN OR Direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 ULN AST (SGOT) and ALT (SGPT) ≤ 2.5 X ULN OR ≤ 5 X ULN for subjects with liver metastases
  * Albumin >2.5 mg/dL
* Coagulation

  * International Normalized Ratio (INR) ≤1.5 X ULN unless subject is receiving therapy as or Prothrombin Time (PT) long as PT or PTT is within therapeutic range of intended use of anticoagulants
  * Activated Partial Thromboplastin Time ≤1.5 X ULN unless subject is receiving (aPTT) anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
* Creatinine clearance should be calculated per institutional standard.
* Negative protein on screening urinalysis
* Female subject of childbearing potential should have a negative serum pregnancy test within 24 hours prior to receiving the first dose of study medication.
* Female subjects of childbearing potential (Section 5.11.2) must be willing to use an adequate method of contraception as outlined in Section 5.11.2 - Contraception, for the course of the study through 120 days after the last dose of study medication. Should a woman become pregnant or suspect she is pregnant while she is participating in this study, she should inform her treating physician immediately.
* Abstinence is acceptable if this is the usual lifestyle and preferred contraception
* Male subjects of reproductive potential (Section 5.11.2) must agree to use an adequate method of contraception as outlined in Section 5.11.2- Contraception, starting with the first dose of study therapy through 120 days after the last dose of study therapy.
* Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.

Exclusion Criteria:

* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
* Has a diagnosis of immunodeficiency including subjects infected with Human Immunodeficiency Virus (HIV).
* Is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
* Has a known history of active TB (Bacillus Tuberculosis).
* Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
* Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.
* Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study.
* If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
* Has a known additional malignancy that is progressing or requires active treatment. -Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
* Lesions suspected to be at higher-risk for bleeding such as bowel involvement with tumor that invades into the bowel wall or involves the intraluminal component of bowel by imaging or direct visualization or central pulmonary lesions.
* Ulcerated skin lesions
* Poorly-controlled hypertension as defined BP > 150/100 mmHg, or SBP > 180 mmHg when DBP < 90 mmHg, on at least 2 repeated determinations on separate days within 3 months prior to study enrollment.
* History within 6 months prior to treatment of myocardial infarction, severe/unstable angina pectoris, CABG, NYHA class III or IV CHF, stroke or TIA.
* History within 3 months prior to treatment of Grade 3-4 GI bleeding/hemorrhage, treatment resistant peptic ulcer disease, erosive esophagitis or gastritis, infectious or inflammatory bowel disease, diverticulitis, pulmonary embolus, or other uncontrolled thromboembolic event.
* Patients who are less than 4 weeks post-op after major surgery.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to pembrolizumab and trebananib including history of allergic reactions to bacterially produced proteins.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Treatment within 30 days prior to enrollment/randomization with strong immune modulators including but not limited to systemic cyclosporine, tacrolimus, sirolimus, mycophenolate mofetil, methotrexate, azathioprine, rapamycin, thalidomide, and lenalidomide.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, interstitial lung disease or active, non-infectious pneumonitis, nephritis, pancreatitis, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis.
* Has an active infection requiring systemic therapy.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
* Patient with ovarian cancer and colorectal cancer who have received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 antibody. Melanoma and renal cell carcinoma patients who received prior anti-PD-1 or ant-PD-L1 or CTLA-4 antibodies are allowed to participate.
* Has received trebananib or another angiopoietin-2 directed therapy (prior treatment with bevacizumab is not an exclusion criteria)
* Has active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
* Has received a live vaccine within 30 days of planned start of study therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2017-08-31 (Actual); Primary Completion 2024-12-13 (Actual); Study Completion 2024-12-13 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicity | 2 years

SECONDARY OUTCOMES:
Objective Response Rate | 2 years
Progression Free Survival | 2 years
Overall Survival | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Hodi, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No